CLINICAL TRIAL: NCT02846675
Title: A Self-control Study: Safety and Efficacy of Autologous Adipose-Derived SVF Cells Delivered Intra-articularly in Patients With Osteoarthritis
Brief Title: Safety and Efficacy of Autologous SVF Cells in Treating Patients With Osteoarthritis
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Shanghai East Hospital (Other)
Responsible Party: Principal Investigator, Yin Feng, Chief Physician, Shanghai East Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DFSC-2014(CR)-03
Record Dates: First submitted 2016-07-25; First posted 2016-07-27 (Estimated); Last update posted 2018-09-11 (Actual); Status verified 2018-09

CONDITIONS: Osteoarthritis
Keywords: SVF; Stromal Vascular Fraction; osteoarthritis(OA); knee; adipose
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- SVF treatment (random knee) (Experimental): A random knee (left or right) of subjects will be treated with autologous SVF.
  Interventions: Biological: autologous SVF
- placebo treatment (the other knee) (Placebo Comparator): The other knee of subjects will be treated with placebo.
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: autologous SVF — SVF will be obtained from lipoaspirates of subjects which will contain more than 5 millions nucleated cells.
  Other Names: Stromal Vascular Fraction
  Arms: SVF treatment (random knee)
Biological: Placebo — a Placebo treatment without SVF cells
  Arms: placebo treatment (the other knee)

SUMMARY:
it's a self-control, double blind study of autologous adipose-derived stromal vascular fraction (SVF) to treat 50 osteoarthritic knees of grade II or III (K-L scale) under IRB-approved protocol in a feasibility and safety study.

DETAILED DESCRIPTION:
The adipose-derived SVF was obtained through disaggregation of lipoaspirate and resuspension of the SVF in 2 ml saline, with at least 50 million nucleated SVF cells and a mean viability of 85%, injected per single knee and the other knee treated with placebo.

Cell suspension and placebo will be injected using ultrasound guidance. Safety and knee function will be evaluated by questionaires monthly and MRI in every three months post-op.

ELIGIBILITY:
Inclusion Criteria:

* Grade II or Grade III osteoarthritis using Kellgren-Lawrence grading scale (K-L Grade) as diagnosed using weight bearing X-ray, physician review, and/or pre-op MRI.
* Study Subjects must have failed a minimum of at least two conservative therapies, spanning a period of at least 3 months.
* Study Subjects must be willing to voluntarily give written Informed Consent to participate in the study and sign the Health Insurance Portability and Accountability Act (HIPAA) authorization before any study procedures are performed.
* Subjects will be in good health (ASA Class I-II) with a BMI < 35.
* Subjects must have continued pain in the knee despite conservative therapies for at least 3 months.
* Subjects with unilateral disease must present with symptomatic knee pain using the WOMAC subscale for pain.
* Subjects must speak, read and understand English.
* Subjects must be reasonably able to return for multiple follow-up visits.

Exclusion Criteria:

* Females who are pregnant or nursing or females of childbearing potential who are unwilling to maintain contraceptive therapy for the duration of the study.
* Life expectancy < 6 months due to concomitant illnesses.
* Exposure to any investigational drug or procedure within 1 month prior to study entry or enrolled in a concurrent study that may confound results of this study.
* Active infectious disease. Patients known to have tested positive for HIV, HTLV, HBV, HCV, CMV (IgM > IgG) and/or syphilis will have an expert consultation as to patient eligibility based on the patient's infectious status
* Any illness which, in the Investigator's judgment, will interfere with the patient's ability to comply with the protocol, compromise patient safety, or interfere with the interpretation of the study results
* Patients on chronic immunosuppressive transplant therapy
* Systolic blood pressure (supine) ≤90 mm Hg or greater than 180mmHg
* Resting heart rate > 100 bpm;
* Known drug or alcohol dependence or any other factors which will interfere with the study conduct or interpretation of the results or who in the opinion of the investigator are not suitable to participate.
* History of cancer (other than non-melanoma skin cancer or in-situ cervical cancer) in the last five years.
* Active clinical infection
* Unwilling and/or not able to give written informed consent.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2014-11-01 (Actual); Primary Completion 2017-07-31 (Actual); Study Completion 2018-01-31 (Actual)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events | 6 months
  Subjects will be monitored for adverse events

SECONDARY OUTCOMES:
Change in Pain Scores on the WOMAC Scale at All Follow-up Visits | 1 month, 2 months, 3 months, 4 months, 5 months, 6 months
  Patients outcomes for pain will be scored through questionaires
Change in Function Scores on the WOMAC Scale at All Follow-up Visits | 1 month, 2 months, 3 months, 4 months, 5 months, 6 months
  Patients outcomes for knee function will be scored through questionaires
Change from baseline in MRI imaging | 3 months & 6 months
  Knee function will be assessed by MRI at three time points: pre-op, 3 months and 6 months post-op

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai East Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Yes